CLINICAL TRIAL: NCT06983496
Title: Pharmacist-Intensivist Collaborative Telehealth for Post-Intensive Care Syndrome in Survivors of Critical Illness: a Pilot Randomized Controlled Trial
Brief Title: Pharmacist-Intensivist Collaborative Telehealth for Post-Intensive Care Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Malcom Randall VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Andrew Franck, Clinical Pharmacy Specialist, Malcom Randall VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202401793
Record Dates: First submitted 2025-04-28; First posted 2025-05-21 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Post Intensive Care Syndrome (PICS)
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth Intervention Group (Experimental): This group will receive the study intervention (i.e. telehealth follow-up appointments at approximately one and three months post-hospital discharge).
  Interventions: Behavioral: Post-ICU Telehealth Follow-up
- Standard of Care Group (No Intervention): This group will receive standard post-ICU care following hospital discharge.

INTERVENTIONS:
Behavioral: Post-ICU Telehealth Follow-up — The post-ICU clinic follow-up will be conducted by a pharmacist via a telehealth visit. A collaborating physician (i.e. intensivist) will provide clinical support and oversight as needed. The appointments will be 30-60 minute telephone/video calls. Participants be assessed for PICS and recommended interventions to improve their care.
  Arms: Telehealth Intervention Group

SUMMARY:
The goal of this pilot randomized controlled trial is to determine if a randomized controlled trial of a collaborative pharmacist-intensivist telehealth follow-up after intensive care unit discharge can feasibly be performed in patients who have survived a critical illness.

The study intervention will be telehealth follow-up appointments provided by clinical pharmacists at approximately one and three months post-hospital discharge. The purpose of the follow-up appointments will be to assess for post-intensive care syndrome and provide recommend interventions aimed at improving recovery

Participants will randomized to receive the study intervention or standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-89 years of age
* Required admission to either medical or surgical ICU
* Respiratory failure requiring invasive mechanical ventilation of at least 24 hours during ICU stay; or ICU stay of at least 7 days
* Anticipated discharge to home after hospitalization
* Consent from patients themselves or a legally authorized representative if necessary

Exclusion Criteria:

* Pregnancy
* Incarceration/Imprisonment
* Life expectancy less than 6 months or enrolled in hospice/palliative care
* Anticipated discharge to skilled nursing facility, medical rehabilitation facility, or other long terms care facility
* Unable to participate in telehealth

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Completion of Post-ICU follow-up | From enrollment to end of follow-up period at seven months
  Percentage of patients completing post-ICU follow-up

SECONDARY OUTCOMES:
Quality of life at 6 months using the Short Form Survey (SF-36) | From enrollment to 7 months
  Medical Outcomes Study (MOS) 36-Item Short Form Health Survey (SF-36). Scores 0-100, higher scores indicating more favorable health state.
Hospital or ICU re-admissions | Enrollment up to 7 months
Emergency department visits | Enrollment up to 7 months
Mortality | within 6 months post-hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Malcom Randall Veterans Affairs Medical Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided